CLINICAL TRIAL: NCT06886126
Title: Phase II Study to Evaluate the Efficacy and Safety of HDM1005 Injection in Obese Nondiabetic Adult Subjects
Brief Title: Phase II Clinical Study of HDM1005 Injection in Obese Adults Without Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HDM1005-202
Record Dates: First submitted 2025-02-12; First posted 2025-03-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- HDM1005 dose cohort 1 QW (Experimental)
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 dose cohort 2 QW (Experimental)
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 dose cohort 3 QW (Experimental)
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 dose cohort 4 QW (Experimental)
  Interventions: Drug: HDM1005 injection or placebo
- placebo QW (Placebo Comparator)
  Interventions: Drug: HDM1005 injection or placebo

INTERVENTIONS:
Drug: HDM1005 injection or placebo — HDM1005 injection subcutaneous injection QW for 22weeks

SUMMARY:
It is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the efficacy and safety of HDM1005 injection in nondiabetic obese adults.

ELIGIBILITY:
Inclusion Criteria:

1. The age of signing ICF was from 18 to 65 years old (including both ends), regardless of gender.

BMI ≥28.0 but <40.0 kg/m2 at screening and randomization 3. Participants reported that they had been under diet and exercise control for 3 months or more before screening, and their weight change (the difference between the maximum body weight and the minimum body weight) in the past 3 months was less than 5%.

(4) fertile female subjects who have taken and agreed to continue to take effective contraceptive measures from 14 days before signing ICF to 60 days after the last dose, and have no plans to give birth and donate eggs; Male subjects signed ICF until 90 days after the last dose, had no fertility plan and sperm donation plan, and agreed to use highly effective contraception.

Exclusion Criteria:

1. Previous diagnosis of type 1, type 2, or any other type of diabetes.
2. History or family history of medullary thyroid carcinoma, C cell hyperplasia, or multiple endocrine neoplasia type 2.
3. According to the investigator's judgment, the subjects have endocrine diseases or histories that affect gastric emptying, may significantly affect body weight, or diseases or conditions that affect the absorption of gastrointestinal nutrients, such as Cushing syndrome, hypothyroidism or hyperthyroidism, bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, and chronic pancreatitis; Or a history of acute pancreatitis or acute gallbladder disease within 3 months before signing ICF.
4. The following cardiovascular and cerebrovascular diseases or conditions occurred within 6 months before randomization:

   1. Unstable angina pectoris;
   2. cardiac insufficiency (New York Heart Association [NYHA] class III or IV);
   3. Myocardial infarction;
   4. Coronary artery bypass grafting or percutaneous coronary intervention;
   5. Severe arrhythmias such as sick sinus syndrome, second or third degree atrioventricular block;
   6. Cerebrovascular accidents, such as cerebral infarction, transient ischemic attack, etc.
5. Hypertension that was not stably controlled at screening: systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg (with stable treatment for at least 30 days if antihypertensive medications were used).
6. Have any malignant tumor within 5 years before signing ICF (except basal cell carcinoma which has received curative treatment and is regarded as cured).
7. Those who had severe infection, severe trauma, or large or medium-sized surgery within 3 months before signing ICF, or planned to undergo surgery during the study (except outpatient surgery).
8. Previous or combined presence or suspicion of depression or other psychiatric disorders or screening PHQ-9 score ≥15.
9. Known intolerance or allergy to any component of the study drug or glucagon-like peptide-1 receptor (GLP-1R) agonist, or a previous history of severe drug allergy.
10. Use of any of the following drugs, products, or treatments within 3 months prior to signing the ICF, including but not limited to:

    A. a drug, product or treatment with weight loss effect b. Medications, products, or treatments that significantly increase body weight
11. Use of hypoglycemic drugs within 3 months before signing ICF.
12. Have participated in any clinical trial within 3 months before signing ICF or within 5 half-lives (whichever is longer) after the last dose of the investigational drug used in the clinical trial (except for those who signed ICF without drug or device intervention).
13. History of addictive drug abuse within 1 year before signing ICF.
14. Any laboratory test during the screening period met the following criteria:

    1. Hemoglobin <100 g/L in women and <110 g/L in men;
    2. alanine aminotransferase >2.5× upper limit of normal (ULN), or aspartate aminotransferase >2.5×ULN, or total bilirubin >1.5×ULN (Gilbert's syndrome subjects with direct bilirubin <ULN can participate in this study);
    3. TG >5.6 mmol/L;
    4. HbA1c ≥6.5%, or fasting plasma glucose ≥7.0 mmol/L or <3.9 mmol/L;
    5. Calcitonin ≥50 ng/L;
    6. Thyroid stimulating hormone >6 mIU/L or <0.4 mIU/L;
    7. serum amylase or lipase >2.0×ULN;
    8. Estimated glomerular filtration rate (eGFR) according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation <60 mL/min/1.73 m2;
    9. Positive test results for active hepatitis B, active hepatitis C, or treponema pallidum antibodies at screening; Antibodies to the human immunodeficiency virus were not negative.
15. Alcohol abuse within 1 year before signing the ICF (i.e. more than 14 standard units per week for men and 7 standard units per week for women, with 1 standard unit containing 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine).
16. Those who donated blood or lost ≥400 mL of total blood within 3 months before signing ICF, or received blood transfusion or used blood products, or planned to donate blood during the study period.
17. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change From Baseline in Body Weight at Week 22 | Baseline, Week 22
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg

SECONDARY OUTCOMES:
Percentage Change From Baseline in Body Weight at Week 4, Week 8, Week 12, Week 16 | Baseline, Week 4, Week 8, Week 12, Week 16
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg
Percentage Change of Participants Achieving Weight Loss ≥ 5% and ≥ 10% at Week 22 | Baseline, Week 22
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg
Change From Baseline in Body Mass Index (BMI) | Baseline, Week 22
  BMI was recorded in kg/m2
Change From Baseline in Waist Circumference | Baseline, Week 22
  Waist Circumference was recorded in cm
Percentage change from baseline in fasting lipid profile (total cholesterol, low density lipoprotein [LDL] cholesterol, high density lipoprotein [HDL] cholesterol, non HDL cholesterol, lipoprotein (a) (Lp[a]), triglycerides) | Baseline, Week 22
  Fasting Lipid Profiles were measured at planned time points.
Change From Baseline in Systolic and Diastolic Blood Pressure | Baseline, Week 22
  Blood Pressure was measured using an automated device
Number of Participants with Clinical Laboratory Abnormalities, and Abnormalities in Vital Signs, Physical Examination and Electrocardiogram and Number of Participants With Treatment Emergent Adverse Events | Baseline to Week 26
  Vital signs (blood pressure, pulse rate, body temperature, respiratory rate), physical examination, ECG and clinical laboratory evaluations (hematology, clinical chemistry, coagulation, urinalysis, calcitonin, serum amylase and lipase)
Pharmacokinetic (PK) Profiles of HDM1005 | Baseline to Week 26
  Antidrug antibodies (ADA) and neutralizing antibody(NAb) profiles of HDM1005

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Doctor, Principal Investigator — Zhongshan Hospital, Shanghai, China
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No